CLINICAL TRIAL: NCT04493307
Title: The Evaluation of Hemostasis by Thromboelastography, Platelet Function Testing, and Biomarker Analysis in Hospitalized COVID-19 Patients
Brief Title: The Evaluation of Hemostasis in Hospitalized COVID-19 Patients
Acronym: TARGET-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: Haemonetics Corporation (Industry); Inflammatory Markers Laboratory (Unknown); Chronolog Corporation (Unknown); Precision Biologics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 1602903
Record Dates: First submitted 2020-06-25; First posted 2020-07-30 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected at study timepoints for the following:
  1. TEG6S with citrated multi-channel and Platelet Mapping cartridges
  2. Platelet aggregation will be assessed using a Chronolog Lumi- Aggregometer
  3. Serum and Plasma Biomarkers of Inflammation/Cytokine Storm, Coagulation,and Ischemia/Organ Injury
  4. Urinary 11-dehydrothromboxane B2
  5. Evaluation of whole blood thrombogenicity using The Total Thrombus- Formation Analysis System (T-TAS)
  6. Genotyping: Genetic variations of single nucleotide polymorphisms (SNPs) related to coagulation, platelet function, immune response and thrombosis related clinical outcomes using SNP microarrays and PCR-based methods.
  7. COVID-19 Antibody Detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Phlebotomy — Serial assessment of hemostasis by blood and urine collection

SUMMARY:
Coronavirus disease 2019 (COVID-19), a viral respiratory illness caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has been shown to predispose patients to thrombotic diseases (venous and arterial) with reported rates in hospitalized patients between 17-40%. The influence of SARS-CoV-2 infection on the coagulation is hypothesized to be regulated by platelet activation, proinflammatory cytokines, endothelial cell injury and stasis. The elevated levels of d-dimer and fibrinogen and clinical signs of organ damage point to a significant hypercoagulable state. The latter induces a high risk for micro-thrombi and multi-organ ischemia. Therefore, early detection and a comprehensive understanding of the influence of the virus on the coagulation and platelet pathways are essential to address this epidemic. It is critical at this time to make all efforts possible to optimize our available technology to care for COVID-19 patients who are at risk for thrombotic disease through appropriate choice, dosing, and laboratory monitoring of antithrombotic therapy.

The investigators hypothesize that COVID-19 is a heightened prothrombotic/hypercoagulability state that can be characterized using platelet function testing and thrombelastography. More information is required to study the effect of COVID-19 on coagulation and platelet pathways to develop effective antithrombotic treatment strategies.

This is a multi-center center, non-interventional study enrolling patients who are COVID-19 positive or who have tested negative showing indication of the disease (high D-dimer and positive lung imaging). The study specific laboratory assessments will be obtained at baseline (closest to time of hospitalization), Day 3, and Day 8 from baseline and at hospital discharge. Laboratory measurements for TEG 6S , platelet aggregation, T-TAS, urinary thromboxane, genotyping, serum and plasma biomarkers will be analyzed . In-hospital and clinical follow-up data will be entered into a COVID registry Patients will be followed for clinical events during hospitalization, and up to 6 months after discharge.

Patients (n=100) hospitalized with at least one of the following will be enrolled.

1. With a confirmed diagnosis of COVID-19 infection using a positive RT- PCR or a positive IgG antibody test prior to or during hospitalization or
2. With a negative COVID-19 RT-PCR test but with symptoms of possible

COVID-19 infection and:

1. an elevated D-dimer and/or
2. positive imaging results showing unilateral or bilateral pneumonia or ground-glass opacity in lungs.

DETAILED DESCRIPTION:
The investigators hypothesize that serial evaluation of (a) intrinsic thrombogenicity measured by thromboelastography (b) platelet activation and aggregation, and (c) selected biomarkers will provide the "blueprint" of individual hemostasis to precisely characterize COVID-19 patients who are at heightened risk for thrombosis or bleeding. The latter will facilitate future efforts to personalize antithrombotic therapy regimens in COVID-19 patients.

Coronavirus disease 2019 (COVID-19), a viral respiratory illness caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has been shown to predispose patients to thrombotic diseases (venous and arterial) with reported rates in hospitalized patients between 17- 40%. The influence of SARS-CoV-2 infection on the coagulation is hypothesized to be regulated by platelet activation, proinflammatory cytokines, endothelial cell injury and stasis.

The elevated levels of d-dimer and fibrinogen and clinical signs of organ damage point to a significant hypercoagulable state. The latter induces a high risk for micro-thrombi and multiorgan ischemia. Therefore, early detection and a comprehensive understanding of the influence of the virus on the coagulation and platelet pathways are essential to address this epidemic. It is critical at this time to make all efforts possible to optimize our available technology to care for COVID-19 patients who are at risk for thrombotic disease through appropriate choice, dosing, and laboratory monitoring of antithrombotic therapy.

Our research group and others have reported a "thrombo-inflammatory" state-a distinct pathophysiological state -of heightened platelet function, hypercoagulability, and inflammation in several cardiovascular disease (CVD) processes. It has been demonstrated that patients with acute respiratory infections are at elevated risk for acute myocardial infarction after influenza (incidence ratio [IR] 6.1, 95% CI 3.9-9.5) and after non-influenza viral illnesses including other coronavirus species (IR 2.8, 95% CI 1.2-6.2). Tantry et al. proposed a mechanistic link between inflammation and heightened thrombogenicity in the presence of unstable CVD state. Furthermore, investigators have hypothesized that this thrombo-inflammatory state becomes even more relevant when patients with CVD and human immunodeficiency virus (HIV) infection undergo percutaneous coronary intervention (PCI).A similar scenario may be present during COVID-19 infection, where evidence of an early myonecrosis may be related to fundamental changes in pathways affecting thrombosis. However, currently, there is no information on how COVID-19 influences hemostasis/thrombosis pathways and subsequent adverse clinical event occurrences.

Cardiovascular comorbidities including hypertension, obesity, high cholesterol, and diabetes mellitus are common in patients with COVID-19 and such patients are at higher risk for morbidity and mortality.12 Furthermore, emerging demographic data in COVID-19 patients shows that incidence and mortality is disproportionately higher in African Americans and Latinos. In a study conducted at Sinai hospital, Lev et al. analyzed a large cohort of racially diverse patients (n=1,172) with CAD or CV risk and demonstrated that sex and race are significantly associated with platelet-fibrin clot strength, a marker of hypercoagulability. Most interesting, AA women had the highest thrombogenicity profile, potentially conferring a highrisk phenotype for thrombotic event occurrence. Furthermore, in a study entitled, "PlateletReactivity in Different Ethnicities" also conducted at Sinai hospital, investigators have demonstrated that Latino and AA races had the highest platelet-fibrin clot strength as compared to Caucasians and others races studied.The latter findings may be described by difference in frequency of a single-nucleotide variant in protease-activated receptor-4 (PAR-4) between AA and Caucasians respectively (63% vs 19%). PAR-4 is an active thrombin receptor on human platelets essential for thrombin-induced platelet activation and has been shown to be more active in African Americans as compared to Caucasians. This evidence may provide a potential mechanistic explanation for racial disparities observed in COVID-19 patients and require further investigation. Hence, investigators will collect a genetic sample to analyze single-nucleotide variant of PAR-4 and other genetic markers related to thrombosis.

Thromboelastography (TEG) is a method for measuring global hemostasis and has been widely used in surgery and anesthesiology, emergency departments, trauma centers, intensive care units,and cardiac catheterization labs for transfusion management, prediction of thrombotic and bleeding events, and choice/adjustment of anticoagulation and antiplatelet therapies. Light transmittance aggregometry (LTA) is a widely used gold standard method for identifying heightened platelet reactivity to various agonists, a marker of thrombotic risk.More common conventional coagulation tests include prothrombin time (PT, INR), partial thromboplastin time (aPTT), fibrinogen, platelet count, and d-dimer. However, these latter tests do not reflect interactions between platelets, endothelium, and fibrinolytic factors and must be used in combination to provide a complete picture of hemostasis status. Unlike these tests, the TEG can assess platelet function, clot strength, and fibrinolysis. Furthermore, The TEG6s Hemostasis Analyzer is a portable, all-in-one cartridge-based system that requires minimal blood sample and minimal sample processing, a potential safety advantage when processing blood samples in COVID-19 patients. Lastly, COVID-19 infection may be associated with acute cardiac injury as indicated by elevation of cardiac biomarkers to > 99th percentile of the upper reference limit, but also electrocardiographic and echocardiographic abnormalities. Cardiac injury is highly prevalent in patients with COVID-19 but may not be an important marker as it occurs after damage has been done. Inosine and hypoxanthine are specific markers of acute cardiac ischemia (ACI) that are measurable within 20 minutes as compared to 4 hours with CKMB and Troponin testing. Investigators believe that this marker may indicate the early presence of micro-thrombi and organ damage. Investigators plan to investigate these novel markers in this trial. Investigators hypothesize that COVID-19 is a heightened prothrombotic/hypercoagulability state that can be characterized using platelet function testing and Thromboelastography. More information is required to study the effect of COVID-19 on coagulation and platelet pathways to develop effective antithrombotic treatment strategies.

The study is a multi-center, non-interventional study involving laboratory testing of blood samples and data collection for a COVID registry using electronic medical records. The study specific laboratory assessments will be obtained at baseline (closest to time of hospitalization), Day 3 and Day 8 from baseline, and at hospital discharge. Patients will be followed for clinical events during hospitalization, and 1 and 6 months after discharge. Patients (n=100) hospitalized at Sinai Hospital of Baltimore and Northwest Hospital with at least one of the following will be enrolled.

1. With a confirmed diagnosis of COVID-19 infection using a positive RT-PCR or a positive IgG antibody test prior to or during hospitalization or,
2. With a negative COVID-19 RT-PCR test but with symptoms of possible COVID-19infection and:

   1. an elevated D-dimer and/or
   2. positive imaging results showing unilateral or bilateral pneumonia or ground glass opacity in lungs.

ELIGIBILITY:
Inclusion Criteria:

* · Confirmed diagnosis of COVID-19 infection using a positive RT-PCR or a positive IgG antibody test prior to or during hospitalization or,

  · With a negative COVID-19 RT-PCR test but with symptoms of possible COVID-19 infection and:
* elevated D-dimer and/or
* positive imaging results showing unilateral or bilateral pneumonia or ground-glass opacity in lungs · The subject or legal authorized representative able to read and sign an informed consent document including authorization permitting release of personal health information approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria:

Subjects will be excluded from entry if ANY of the criteria listed below are met:

* Less than 3 years of age
* Subject is pregnant
* Active treatment for cancer
* History of long-term use of immunosuppressive agents
* History of severe chronic respiratory disease and requirement for long-term oxygen therapy
* Patients undergoing hemodialysis or peritoneal dialysis
* Patients on full dose anticoagulant at the time of enrollment
* Any condition unsuitable for the study as determined by investigators

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study's intended population is inclusive of both genders (males and females), aged 3 years and older, and all racial and ethnic groups.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of Hypercoagulability as measured by thromboelastography measured by TEG and platelet aggregation. | up to day 8
  Frequency of Hypercoagulability as measured by point-of-care thromboelastography (TEG6s)

SECONDARY OUTCOMES:
Frequency of High Platelet Reactivity (HPR) | up to day 8
  Incidence of High Platelet Reactivity as measured by platelet aggregation and TEG6s
Frequency of thrombo-inflammatory syndrome | up to day 8
  Frequency of thrombo -inflammatory syndrome as determined by D-Dimer and TEG6s
Correlation between TEG6s parameters and clinical outcomes | through study completion, an average of 6 months
  Correlation between TEG6s parameters and clinical outcomes (thrombotic and bleeding events, need for ventilation, death)
Correlation between HPR and clinical outcomes | through study completion, an average of 6 months
  Correlation between HPR and clinical outcomes (thrombotic and bleeding events, need for ventilation, death)
Determine response to anticoagulation therapy | up to day 8
  Determine response to anticoagulation therapy by calculating change in R-value (CK -CKH)
Determine level of platelet aggregation | up to day 8
  Determine level of platelet aggregation by impedance aggregometry
Determine level of platelet aggregation | up to day 8
  Determine percent platelet aggregation by TEG-6S platelet Mapping assay
Determine platelet thrombi and fibrin rich platelet thrombus Area Under the Curve | up to day 8
  Determine platelet thrombi and fibrin rich platelet thrombus Area Under the Curve using TTAS analyzer
Determine short and long IgG, IgM and IgG antibody levels | up to day 6 months
  Determine short and long IgG, IgM and IgG antibody levels against using multiple specimen types (saliva, whole blood, serum, plasma, urine)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurbel PA, Bliden KP, Levy JH, Walia N, Rapista N, Cho A, Jerjian C, Tantry US. Thrombogenicity markers for early diagnosis and prognosis in COVID-19: a change from the current paradigm? Blood Coagul Fibrinolysis. 2021 Dec 1;32(8):544-549. doi: 10.1097/MBC.0000000000001069. PMID 34369413